CLINICAL TRIAL: NCT05739929
Title: Colchicine Protective Effect in Patients Undergoing Elective Percutaneous Coronary Intervention (COLCHICINE-PROTECT) A Randomized, Placebo-controlled, Double-blind Clinical Trial
Brief Title: Colchicine Protective Effect in Patients Undergoing Percutaneous Coronary Intervention (COLCHICINE-PROTECT)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Shafie Ammar, Assistant Lecturer of Cardiology, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 120-2022
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Acute Coronary Syndrome; Percutaneous Coronary Intervention; Colchicine; Myocardial Injury; Inflammation; Myocardial Infarction; No Reflow
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Inflammation; Myocardial Infarction | interventions — Colchicine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Active Comparator): 0.5 mg colchicine tablets twice daily 72 to 48 hours before planned PCI
  Interventions: Drug: Colchicine 0.5 MG Oral Tablet
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 MG Oral Tablet — 0.5 mg colchicine tablets twice daily.
  Other Names: Colcrys; Gloperba; Mitigare
  Arms: Colchicine
Drug: Placebo — Placebo tablets twice daily
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the colchicine protective effect in patients undergoing Percutaneous Coronary Intervention (PCI). The main question it aims to answer is: does initiating colchicine before planned PCI will reduce post-procedural myocardial injury? Half of the participants will receive colchicine, while the other half will receive a placebo.

DETAILED DESCRIPTION:
Inflammation in the setting of PCI is associated with endothelial dysfunction and microvascular obstruction and remains an independent predictor of subsequent major adverse cardiovascular events (MACE) even in the contemporary era of second-generation drug-eluting stents (DES). Inflammation also increases the risk of PCI-related myocardial injury, which is associated with long-term all-cause mortality.

Colchicine is an inexpensive, orally administered, potent anti-inflammatory medication. Recent major trials showed that using low-dose colchicine on top of GDMT reduces cardiovascular events in patients with either chronic coronary syndrome (CCS) or acute Myocardial infarction (MI).

A recent meta-analysis showed that using colchicine in the setting of PCI also reduces cardiovascular events, however, the optimal regimen to subside PCI-associated inflammation is still not clear.

Our aims are

1. Evaluation of colchicine efficacy in protecting against PCI myocardial injury. Our hypothesis is that initiating colchicine 0.5 mg twice daily 72 to 48 hours before planned PCI in CCS patients will decrease PCI-related myocardial injury.
2. Evaluation of colchicine efficacy in preventing PCI-associated inflammation. Our hypothesis is that colchicine will subside post-PCI rise in high sensitive C-Reactive-Protein (hs-CRP).
3. Evaluation of colchicine efficacy in preventing no-reflow phenomenon. Our hypothesis is that colchicine will decrease no reflow phenomenon in CCS patients undergoing PCI.
4. Evaluation of colchicine efficacy in preventing PCI-related (type 4a) MI per the 4th Universal Definition. Our hypothesis is that colchicine will decrease PCI-related (type 4a) MI in CCS patients undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Coronary Syndrome (CCS) participants referred for PCI.
* Acute Coronary Syndrome (ACS) participants who are medically treated or undergoing revascularization for non-culprit lesions will be included if their troponin I and hs-CRP returned back to normal baseline

Exclusion Criteria:

* Acute Coronary Syndrome (ACS) participants.
* Chronic kidney disease (glomerular filltration rate <30 ml/ min).
* Participants with history of cirrhosis.
* Participants on systemic immunosuppressive or corticosteroid therapy.
* Active malignancy or infection.
* Elevated troponin I.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
PCI related myocardial injury | 6 hours after PCI
  Number of Participants with peak post-procedure Troponin I above the upper reference limit in participants with normal baseline cardiac biomarkers

SECONDARY OUTCOMES:
PCI associated inflammation | 6 hours after PCI
  Post PCI hs-CRP
No reflow phenomenon | During the PCI procedure
  Defined as Thrombolysis in Myocardial Infarction (TIMI) flow grade of less than 3.
PCI-related (type 4a) Myocardial Infarction (MI) | 6 hours after PCI
  According to the 4th Universal Definition of MI

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Ammar, MD, MSc, Principal Investigator — Helwan University, Faculty of Medicine
Locations (1):
- Helwan University Hospital, Helwan, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
"De-identified individual participant data collected during the COLCHICINE-PROTECT trial will be shared at 2 years after article publication with no end date. These data will be available to researchers who provide a methodologically sound proposal for the purposes of achieving specific aims outlined in that proposal. Proposals should be directed to Mohammed A Ammar via email (mohammed.ahmed5@med.helwan.edu.eg) and will be reviewed by the COLCHICINE-PROTECT study management committee. Requests to access data to undertake hypothesis-driven research will not be unreasonably withheld. To gain access, data requesters will need to sign a data access agreement and to confirm that data will only be used for the agreed purpose for which access was granted."
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: at 2 years after article publication with no end date.
Access Criteria: These data will be available to researchers who provide a methodologically sound proposal for the purposes of achieving specific aims outlined in that proposal.
  Proposals should be directed to Mohammed A Ammar via email (mohammed.ahmed5@med.helwan.edu.eg) and will be reviewed by the COLCHICINE-PROTECT study management committee. Requests to access data to undertake hypothesis-driven research will not be unreasonably withheld. To gain access, data requesters will need to sign a data access agreement and to confirm that data will only be used for the agreed purpose for which access was granted."

REFERENCES:
- [Background] Kwaijtaal M, van Diest R, Bar FW, van der Ven AJ, Bruggeman CA, de Baets MH, Appels A. Inflammatory markers predict late cardiac events in patients who are exhausted after percutaneous coronary intervention. Atherosclerosis. 2005 Oct;182(2):341-8. doi: 10.1016/j.atherosclerosis.2005.02.022. Epub 2005 Mar 24. PMID 16159607
- [Background] Writing Committee Members; Lawton JS, Tamis-Holland JE, Bangalore S, Bates ER, Beckie TM, Bischoff JM, Bittl JA, Cohen MG, DiMaio JM, Don CW, Fremes SE, Gaudino MF, Goldberger ZD, Grant MC, Jaswal JB, Kurlansky PA, Mehran R, Metkus TS Jr, Nnacheta LC, Rao SV, Sellke FW, Sharma G, Yong CM, Zwischenberger BA. 2021 ACC/AHA/SCAI Guideline for Coronary Artery Revascularization: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2022 Jan 18;79(2):e21-e129. doi: 10.1016/j.jacc.2021.09.006. Epub 2021 Dec 9. PMID 34895950
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Novack V, Pencina M, Cohen DJ, Kleiman NS, Yen CH, Saucedo JF, Berger PB, Cutlip DE. Troponin criteria for myocardial infarction after percutaneous coronary intervention. Arch Intern Med. 2012 Mar 26;172(6):502-8. doi: 10.1001/archinternmed.2011.2275. Epub 2012 Feb 27. PMID 22371874
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Angelantonio ED, Franco OH, Halvorsen S, Richard Hobbs FD, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice: Developed by the Task Force for cardiovascular disease prevention in clinical practice with representatives of the European Society of Cardiology and 12 medical societies With the special contribution of the European Association of Preventive Cardiology (EAPC). Rev Esp Cardiol (Engl Ed). 2022 May;75(5):429. doi: 10.1016/j.rec.2022.04.003. No abstract available. English, Spanish. PMID 35525570
- [Result] Cole J, Htun N, Lew R, Freilich M, Quinn S, Layland J. Colchicine to Prevent Periprocedural Myocardial Injury in Percutaneous Coronary Intervention: The COPE-PCI Pilot Trial. Circ Cardiovasc Interv. 2021 May;14(5):e009992. doi: 10.1161/CIRCINTERVENTIONS.120.009992. Epub 2021 May 18. PMID 34003667
- [Result] Fu C, Wang B. Colchicine administration for percutaneous coronary intervention: A meta-analysis of randomized controlled trials. Am J Emerg Med. 2021 Aug;46:121-125. doi: 10.1016/j.ajem.2021.02.039. Epub 2021 Feb 22. PMID 33744748
- [Result] Shah B, Pillinger M, Zhong H, Cronstein B, Xia Y, Lorin JD, Smilowitz NR, Feit F, Ratnapala N, Keller NM, Katz SD. Effects of Acute Colchicine Administration Prior to Percutaneous Coronary Intervention: COLCHICINE-PCI Randomized Trial. Circ Cardiovasc Interv. 2020 Apr;13(4):e008717. doi: 10.1161/CIRCINTERVENTIONS.119.008717. Epub 2020 Apr 16. PMID 32295417
- [Result] Hosseini SH, Talasaz AH, Alidoosti M, Tajdini M, Van Tassell BW, Etesamifard N, Kakavand H, Jalali A, Aghakouchakzadeh M, Gheymati A, Sadeghian M, Jenab Y. Preprocedural Colchicine in Patients With Acute ST-elevation Myocardial Infarction Undergoing Percutaneous Coronary Intervention: A Randomized Controlled Trial (PodCAST-PCI). J Cardiovasc Pharmacol. 2022 Oct 1;80(4):592-599. doi: 10.1097/FJC.0000000000001317. PMID 35881907
- [Result] Maron DJ, Hochman JS, Reynolds HR, Bangalore S, O'Brien SM, Boden WE, Chaitman BR, Senior R, Lopez-Sendon J, Alexander KP, Lopes RD, Shaw LJ, Berger JS, Newman JD, Sidhu MS, Goodman SG, Ruzyllo W, Gosselin G, Maggioni AP, White HD, Bhargava B, Min JK, Mancini GBJ, Berman DS, Picard MH, Kwong RY, Ali ZA, Mark DB, Spertus JA, Krishnan MN, Elghamaz A, Moorthy N, Hueb WA, Demkow M, Mavromatis K, Bockeria O, Peteiro J, Miller TD, Szwed H, Doerr R, Keltai M, Selvanayagam JB, Steg PG, Held C, Kohsaka S, Mavromichalis S, Kirby R, Jeffries NO, Harrell FE Jr, Rockhold FW, Broderick S, Ferguson TB Jr, Williams DO, Harrington RA, Stone GW, Rosenberg Y; ISCHEMIA Research Group. Initial Invasive or Conservative Strategy for Stable Coronary Disease. N Engl J Med. 2020 Apr 9;382(15):1395-1407. doi: 10.1056/NEJMoa1915922. Epub 2020 Mar 30. PMID 32227755
- [Result] Munk PS, Breland UM, Aukrust P, Skadberg O, Ueland T, Larsen AI. Inflammatory response to percutaneous coronary intervention in stable coronary artery disease. J Thromb Thrombolysis. 2011 Jan;31(1):92-8. doi: 10.1007/s11239-010-0471-7. PMID 20373128
- [Result] Nidorf SM, Fiolet ATL, Mosterd A, Eikelboom JW, Schut A, Opstal TSJ, The SHK, Xu XF, Ireland MA, Lenderink T, Latchem D, Hoogslag P, Jerzewski A, Nierop P, Whelan A, Hendriks R, Swart H, Schaap J, Kuijper AFM, van Hessen MWJ, Saklani P, Tan I, Thompson AG, Morton A, Judkins C, Bax WA, Dirksen M, Alings M, Hankey GJ, Budgeon CA, Tijssen JGP, Cornel JH, Thompson PL; LoDoCo2 Trial Investigators. Colchicine in Patients with Chronic Coronary Disease. N Engl J Med. 2020 Nov 5;383(19):1838-1847. doi: 10.1056/NEJMoa2021372. Epub 2020 Aug 31. PMID 32865380
- [Result] Tardif JC, Kouz S, Waters DD, Bertrand OF, Diaz R, Maggioni AP, Pinto FJ, Ibrahim R, Gamra H, Kiwan GS, Berry C, Lopez-Sendon J, Ostadal P, Koenig W, Angoulvant D, Gregoire JC, Lavoie MA, Dube MP, Rhainds D, Provencher M, Blondeau L, Orfanos A, L'Allier PL, Guertin MC, Roubille F. Efficacy and Safety of Low-Dose Colchicine after Myocardial Infarction. N Engl J Med. 2019 Dec 26;381(26):2497-2505. doi: 10.1056/NEJMoa1912388. Epub 2019 Nov 16. PMID 31733140